CLINICAL TRIAL: NCT05603845
Title: Patient-Reported OUTcomes of Benralizumab in Real-World Use in Severe EosiNophilic Asthma Patients Multicountry, Multicenter, Observational, Prospective, Primary Data, Real-world Settings
Brief Title: Patient-Reported OUTcomes of Benralizumab in Real-World Use in Severe EosiNophilic Asthma Patients
Acronym: iOUTRUN
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00113
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Severe Asthma
Keywords: Severe Asthma; Benralizumab; Eosinophilic asthma; Patient reported outcomes
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to generate real-world data on the characteristics of patients receiving benralizumab to assess early PRO parameters as well as long-term treatment effects in the Gulf cooperative council (Kingdom of Saudi Arabia, Kuwait, United Arab Emirates, Oman, and Qatar), Latin America (Brazil, Argentina, and Colombia), and India. It is anticipated that the data generated will provide practical, patient-focused real-world evidence and enhance communications between patients and physicians in an objective and structured manner to ensure better disease control in patients under benralizumab treatment.

DETAILED DESCRIPTION:
This is a multi-country, multi-center, observational, prospective study involving primary data collection within real-world pulmonary care settings for patients who receive benralizumab treatment for severe uncontrolled eosinophilic asthma.The decision by the physician to start benralizumab is made independently from study inclusion and patient informed consent. Patients will receive benralizumab injections according to the local label in the participating countries (Brazil, Argentina, Colombia, India, and the Gulf cooperative council, including the Kingdom of Saudi Arabia, United Arab Emirates, Kuwait, Oman, and Qatar). No study drug will be provided as part of the study. The entire study period duration will be 56 weeks for each subject. The study is anticipated to run for approximately 18 months and is not anticipated to exceed 24 months. A database soft lock is planned at the end of the initial 8-week period of the study, and one combined descriptive and analytical interim analysis will be performed when 50% of the enrolled subjects complete the 8-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 years or older with a physician's confirmed diagnosis of severe eosinophilic, uncontrolled asthma.
2. Severe uncontrolled eosinophilic asthma requiring high-dose* inhaled corticosteroid plus long-acting β adrenoceptor agonist as maintenance treatment.
3. Patients who have been prescribed but not yet initiated treatment with benralizumab (Fasenra®) according to local approved prescribing information prior to signed informed consent.
4. Provision of the signed written informed consent form (ICF) indicating that they understand the purpose of the study and procedures required for participation.
5. Patients must be able and willing to read and comprehend written instructions and complete the paper PRO questionnaires required by the protocol.

Exclusion Criteria:

1. Clinically important pulmonary diseases other than asthma including chronic obstructive pulmonary disease (as the main diagnosis), bronchiectasis, idiopathic pulmonary fibrosis, pulmonary hypertension, alpha-1-antitrypsin-deficiency, and malignancy of any kind (NB: the following conditions are permitted: nasal polyposis, allergic rhinitis, atopic dermatitis, non-idiopathic pulmonary fibrosis).
2. Currently enrolled in an interventional clinical study except patients being in parallel documented in a national asthma registry
3. An acute or chronic condition that, in the investigator's opinion, would limit the patients' ability to complete questionnaires or participate in this study or impact the interpretations of results.
4. Concurrent biologics for asthma are not allowed. Acceptable wash-out periods for other asthma biologics: ≥30 days from the last dose of the previous biologic.
5. Women who are currently pregnant, breastfeeding, or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will recruit 410 adult patients with confirmed severe eosinophilic asthma who meet all inclusion criteria and none of the exclusion criteria in 9 countries as described above.
  Approximately 6-8 hospitals per country will participate in the study which have previous experience with biologic treatment, can initiate treatment with benralizumab, and have a good oversight on the severe asthma population.
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Asthma Control Questionnaire (ACQ-6) | 8 weeks
  The changes from baseline in Asthma Control Questionnaire (ACQ-6) score at eight weeks of benralizumab treatment.
  Minimum Value - '0' Maximum Value - '6' The lower the value better is the outcome

SECONDARY OUTCOMES:
Changes from baseline in Asthma Control Questionnaire (ACQ-6) | 56 weeks
  The changes from baseline in Asthma Control Questionnaire (ACQ-6) score at 1, 2, 3, 4, 24, and 56 weeks of benralizumab treatment.
  Minimum Value - '0' Maximum Value - '6' The lower the value better is the outcome.
Percentage of patients with a total score improvement with regards to Minimal clinically important difference in ACQ-6 (Asthma controlled questionnaire) | 56 weeks
  Percentage of patients with a total score improvement of ≥ 0.5 points (minimal clinically important difference [MCID]) in ACQ-6 (Asthma controlled questionnaire) at 1, 2, 3, 4, 8, 24, and 56 weeks of receiving benralizumab compared to baseline Minimum Value - '0' Maximum Value - '6' The lower the value better is the outcome.
Percentage of patients based on their Asthma control using ACQ-6 | 56 weeks
  Percentage of patients with well-controlled asthma (ACQ-6 ≤ 0.75), partly controlled asthma (ACQ-6 between >0.75 and <1.5), and uncontrolled asthma (ACQ-6 ≥ 1.5) at baseline and at 1, 2, 3, 4, 8, 24, and 56 weeks of benralizumab treatment Minimum Value - '0' Maximum Value - '6' The lower the value better is the outcome.
Patient global impression of change (PGI-C) response | 56 weeks
  The patient global impression of change (PGI-C) response at 1, 2, 3, 4, 8, 24, and 56 weeks of benralizumab treatment Minimum Value - '1' Maximum Value - '7' The lower the value better is the outcome
Patient global impression of severity (PGI-S) response | 56 weeks
  The patient global impression of severity (PGI-S) response at 0, 1, 2, 3, 4, 8, 24, and 56 weeks of benralizumab treatment Minimum Value - '1' Maximum Value - '6' The lower the value better is the outcome
Pre-bronchodilator forced expiratory volume in the first second (FEV1) | 56 weeks
  Changes in the Pre-bronchodilator forced expiratory volume in the first second (Pre BD - FEV1) Unit - "ml' It will measure the change value - The higher the better
Change from baseline of the patient-reported nasal polyposis symptoms | 56 weeks
  Change from baseline using the visual analog scale (VAS) for the following parameters
  1. Loss of smell
  2. Nasal blockage/nasal Congestion
  3. Difficulty with sleeping due to nasal symptoms
  4. Headache/Pressure on face
  Minimum Value - '1' Maximum Value - '10' The lower the value better is the outcome.
Pre-bronchodilator forced vital capacity (FVC) changes | 56 weeks
  Change in the pre-BD Forced vital capacity (FVC) changes Unit - "ml' It will measure the change value - The higher the better
Percentage of patients who achieved 100 ml improvement in their lung function | 56 Weeks
  Percentage of patients who achieved 100 ml improvement in their lung function (Pre BD - FEV1) This will be measured as '%' More the value better is the outcome

CONTACTS AND LOCATIONS:
Locations (24):
- Colombia (4):
  - Research Site, Bogotá
  - Research Site, Bucaramanga
  - Research Site, Ibagué
  - Research Site, Pereira
- Dominican Republic (2):
  - Research Site, Santiago de los Caballeros
  - Research Site, Santo Domingo
- India (10):
  - Research Site, Ahmedabad
  - Research Site, Ajmer
  - Research Site, Chennai
  - Research Site, Delhi
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Kolkata
  - Research Site, Pune
  - Research Site, Secundrabad
  - Research Site, Vadodara
- Research Site, Sabah Al Salem, Kuwait
- Research Site, Muscat, Oman
- Research Site, Doha, Qatar
- Saudi Arabia (2):
  - Research Site, Jeddah
  - Research Site, Riyadh
- United Arab Emirates (3):
  - Research Site, Abu Dhabi
  - Research Site, Al Ain City
  - Research Site, Dubai

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home